CLINICAL TRIAL: NCT07023224
Title: Adaptation Of The Parkinson's Disease Dyskinesia Questionnaire Into Turkish And Its Validity And Reliability In Parkinson's Patient
Brief Title: Reliability and Validity Study of the Turkish Version of the Parkinson's Disease Dyskinesia Scale (PDYS-26)
Status: Recruiting | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Irem Tepe Bark, Principal Investigator, Izmir Bakircay University
Other Study IDs: IZBU-FTR-ITB-01
Record Dates: First submitted 2025-05-28; First posted 2025-06-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Parkinson Disease; Dyskinesias; Quality of Life
Keywords: Parkinson's disease; Dyskinesia; Parkinson's Disease Dyskinesia Scale
MeSH Terms: conditions — Parkinson Disease; Dyskinesias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson Patients with Dyskinesia: Parkinson's disease patients with a Unified Parkinson's Disease Rating Scale (UPDRS) dyskinesia score of ≥1. Participants must meet the inclusion criteria and provide informed consent.
  Interventions: Other: Turkish version of the Parkinson's Disease Dyskinesia Scale (PDYS-26)

INTERVENTIONS:
Other: Turkish version of the Parkinson's Disease Dyskinesia Scale (PDYS-26) — The Turkish adaptation of the Parkinson's Disease Dyskinesia Scale (PDYS-26) is administered to individuals diagnosed with Parkinson's disease who have a dyskinesia score of ≥1 based on the Unified Parkinson's Disease Rating Scale (UPDRS) dyskinesia item. The scale is used to evaluate dyskinesia severity and assess its clinical applicability in Turkish-speaking populations.

SUMMARY:
The aim of this methodological study was to investigate the Turkish validity and reliability of the Parkinson's Disease Dyskinesia Scale (PDYS-26).The scale evaluates choreic dyskinesia.Measures the impact of dyskinesia on activities of daily living in patients with Parkinson's disease.

Hypotheses of the Study:

* Parkinson's Disease Dyskinesia Scale (PDYS-26) is reliable in Turkish.
* Parkinson's Disease Dyskinesia Scale (PDYS-26) is valid in Turkish.

To determine the validity of dyskinesia;

* Tampa Kinesiophobia Scale,
* Mini BesTest,
* Activity Specific Balance Safety Scale (ABC) and
* Parkinson's Disease Questionnaire-39 will be evaluated.

DETAILED DESCRIPTION:
In Parkinson's disease, a neurodegenerative disorder affecting the peripheral and central nervous system, dyskinesia is a common symptom that occurs as disease processes progress and leads to disability. The term dyskinesia is a general term that covers many movement disorders. In general, it can be defined as mild to severe abnormal and involuntary muscle movements. In individuals with Parkinson's disease, it is a natural consequence of the neurodegenerative process and a motor complication of the gold standard L-dopa. Assessment of dyskinesia in Parkinson's patients is important for the implementation of appropriate medical, surgical and rehabilitation protocols. There are few scales and patient diaries that clinically assess the effect of interventions for dyskinesia. At the same time, there are deficiencies related to the reliability and validity studies of these existing scales in different languages. Therefore, limitations may arise in the assessment of dyskinesia. For this purpose, our study aims to investigate the reliability and validity of the Parkinson's Disease Dyskinesia Scale (PDYS-26) in Turkish in patients diagnosed with 130 idiopathic Parkinson's patients.In the study, the Parkinson's Disease Dyskinesia Scale (PDYS-26) will be translated into Turkish with the "back translation" method and will be finalized after the approval of the commission consisting of relevant health professionals. The final version of the scale will be applied to Parkinson's patients. To determine the validity of dyskinesia; Tampa Kinesiophobia Scale, Mini BesTest Activity Specific Balance Safety Scale (ABC) and Parkinson's Disease Questionnaire-39 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with idiopathic Parkinson's disease
* H&Y stage 1-3
* UPDRS dyskinesia item score ≥1
* Accepting to participate in the study

Exclusion Criteria:

* Diagnosis of atypical-secondary parkinsonism
* Severe musculoskeletal, neurological and/or cardiopulmonary problems that may affect the results of the assessment
* Mini Mental State Examination score < 24

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study was planned as a methodological research. For this purpose, Parkinson's disease patients who applied to Izmir Çiğli Training and Research Hospital Neurology Outpatient Clinic and met the inclusion criteria will be included in the study. Written informed consent will be obtained from individuals who agree to participate in the study. Based on the commonly recommended participant-to-item ratio in validity and reliability studies (typically 5 to 10 participants per item), the sample size was determined as five times the number of items in the 26-item PDYS-26 scale, and a total of 130 patients with Parkinson's disease were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
(PDYS-26) | Baseline (Day 1) and 7 days post-baseline (Day 8)
  Turkish version of Parkinson's Disease Dyskinesia Scale: It is a questionnaire that assesses the impact of dyskinesia on activities of daily living. It consists of 26 items. A higher score indicates greater impact.It is considered a consistent, reliable, and valid measure. It is easy to complete and has a short administration time.

OTHER OUTCOMES:
Tampa Kinesiophobia Scale | Baseline (Day 1)
  Tampa Kinesiophobia Scale: It consists of 17 items that assess avoidance of movement due to a history of injury or pain.
  The minimum score is 17 and the maximum score is 68; a score of 37 or above indicates a high level of kinesiophobia.
  A 4-point Likert scale is used to evaluate the responses (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree).
(Mini-BesTest) | Baseline (Day 1)
  Mini BesTest Balance Scale: It is one of the clinical tests used to assess gait and balance. It consists of 4 subcomponents: anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait, with a total of 14 items. A higher score indicates better function.
(ABC) | Baseline (Day 1)
  Activity Specific Balance Safety Scale: It evaluates the individual's perceived level of confidence during balance-related activities of daily living.
  The level of confidence is assessed by the evaluator through 16 items directly asked to the individual, with scores ranging from 0% (no confidence) to 100% (complete confidence).
  A total score between 0 and 49 indicates a low functional level, 50 to 80 indicates a moderate functional level, and 81 to 100 indicates a high functional level.
(PDQ-39) | Baseline (Day 1)
  Parkinson's Disease Questionnaire-39: It is one of the most commonly used scales for assessing quality of life in individuals with Parkinson's disease.
  It evaluates the impact of Parkinson's disease on quality of life over the past month. Lower total scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gulbın Ergın, PT, PhD, Principal Investigator — Izmir Bakircay Univercity
Locations (2):
- Turkey (Türkiye) (2):
  - Bakirçay University Çiğli Regional Education Hospital, Izmir, İ̇zmi̇r
  - Izmir Bakırçay Univercity, Izmir

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared beyond the research team due to ethical and confidentiality considerations.

REFERENCES:
- [Background] Katzenschlager R, Schrag A, Evans A, Manson A, Carroll CB, Ottaviani D, Lees AJ, Hobart J. Quantifying the impact of dyskinesias in PD: the PDYS-26: a patient-based outcome measure. Neurology. 2007 Aug 7;69(6):555-63. doi: 10.1212/01.wnl.0000266669.18308.af. PMID 17679674
- See also: The original publication of the scale that is the subject of the Turkish adaptation study — https://pubmed.ncbi.nlm.nih.gov/17679674/